CLINICAL TRIAL: NCT05134220
Title: Study of Serum Calcium and Phosphorus Level in Chronic Kidney Disease Patients With Acute Coronary Syndrome
Brief Title: Electrolytes in Chronic Kidney Disease Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Youssif, Principal Investigator, Sohag University
Other Study IDs: Electrolytes
Record Dates: First submitted 2021-11-06; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Kidney Disease (CKD) patients with acute coronary syndrome: The CKD patients with or without dialysis who admitted to coronary care unit with chest pain consistent with ACS with any of following features :
  1. Electrocardiogram (ECG) changes:
     * ST elevation.
     * ST depression.
     * T wave inversion.
     * recent left bundle branch block.
  2. Troponin elevation.
  Interventions: Diagnostic Test: Serum Calcium
- Chronic Kidney Disease (CKD) patients without acute coronary syndrome: The CKD patient with or without dialysis with no previous history of ACS.
  Interventions: Diagnostic Test: Serum Calcium

INTERVENTIONS:
Diagnostic Test: Serum Calcium — * Serum calcium level.
  * Serum phosphorus level. will be measured to all study population
  Other Names: serum Phosphorus

SUMMARY:
Study of serum calcium and phosphorus level in chronic kidney disease patients and its relation to occurrence of acute coronary syndrome in them.

DETAILED DESCRIPTION:
Prospective study to :

1. find the relation between electrolytes disturbance and renal diseases
2. the effect of electrolyte abnormalities on atherosclerosis
3. prevalence of acute coronary syndrome in patients with chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* 1-The CKD patients with or without dialysis who admitted to coronary care unit with chest pain consistent with ACS with any of following features :

  a- Electrocardiogram (ECG) changes:
* ST elevation.
* ST depression.
* T wave inversion.
* recent left bundle branch block.

  b- Troponin T elevation.

  2-The CKD patient with or without dialysis with no previous history of ACS.

Exclusion Criteria:

1. Patients who were diagnosed with primary hyperparathyroidism.
2. Acute Kidney injury (AKI) which is defined as any of the following:(KDIGO2012)

   * Increase in S.Cr by ≥ 0.3 mg/dl (≥ 26.5 μmol/l) within 48hours; or
   * Increase in S.Cr to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days;or
   * Urine volume <0.5 ml/kg/h for 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: two groups :
  1. CKD patients with and without dialysis who admitted to Sohag university hospital with acute coronary syndrome
  2. CKD patients with and without dialysis who admitted to Sohag university hospital with no previous or current history of acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Chronic kidney disease hospitalization | from the day of admission to the day of discharge through study completion, an average of 28 weeks, in sohag university hospital
  The CKD patient with and without acute coronary syndrome and estimated hazard ratios (HR) by use of multivariable Cox regression models.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

REFERENCES:
- [Background] Block GA, Hulbert-Shearon TE, Levin NW, Port FK. Association of serum phosphorus and calcium x phosphate product with mortality risk in chronic hemodialysis patients: a national study. Am J Kidney Dis. 1998 Apr;31(4):607-17. doi: 10.1053/ajkd.1998.v31.pm9531176.